CLINICAL TRIAL: NCT05211219
Title: The Role of Probiotics in Preventing Dysbiosis in Periodontal Disease
Brief Title: The Role of Probiotics in Periodontal Disease
Acronym: tropipd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurdan Ozmeric, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/2020-18; 6268 (Other Grant/Funding Number: Gazi University Project of Science Investigation)
Record Dates: First submitted 2021-11-26; First posted 2022-01-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases
Keywords: Periodontal disease; Probiotics; Prebiotics
MeSH Terms: conditions — Periodontal Diseases | interventions — Probiotics; Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics (Experimental): The probiotics group was advised to consume a chewable tablet once a day in 14 days.
  Interventions: Dietary Supplement: Probiotics
- Kefir (Experimental): The kefir group was advised to consume kefir as a liquid once a day in 14 days.
  Interventions: Dietary Supplement: AOÇ Kefir
- Control (Other): the control group was advised without additional food supplements.
  Interventions: Other: Food without additional food supplements

INTERVENTIONS:
Dietary Supplement: Probiotics — According to the groups, they were involved simultaneously with the treatment, kefir group was advised to consume kefir as a liquid once a day in 14 days; the probiotics group was advised to consume as a chewable tablet once a day in 14 days; the control group was advised without additional food supplements.
  Other Names: Probest Defense
  Arms: Probiotics
Dietary Supplement: AOÇ Kefir — AOÇ Kefir
  Arms: Kefir
Other: Food without additional food supplements — Food without additional food supplements
  Arms: Control

SUMMARY:
In this randomized controlled trial, it was aimed to evaluate the effect of probiotics (chewable tablets) and kefir consumption in the initial periodontal treatment of periodontitis patients on the change of oral microbiota and treatment. In this clinical trial, 36 systemically healthy volunteers who were diagnosed with periodontitis who were admitted to Gazi University Faculty of Dentistry, Department of Periodontology were included. Besides the inclusion criteria, the nutritional habits of the patients were evaluated by questionnaire. For diagnosis, plaque index, gingival index, bleeding on probing, periodontal probing depth and clinical attachment level were examined. Patients were randomly divided into 3 groups; probiotic, kefir and control group. Following the periodontal diagnosis, clinical index records of the patients and subgingival microbial samples were obtained. The supragingival plaque sample was removed and the subgingival microbial dental plaque sample was gently taken with a sterile Gracey curette. In the same session, periodontal initial treatment was started. According to the groups, they were involved simultaneously with the treatment, kefir group was advised to consume kefir as a liquid once a day in 14 days; probiotics group was advised to consume as a chewable tablet once a day in 14 days; the control group was advised without additional food supplements. Periodontal indexes were repeated in the 1st and 3rd months. Subgingival plaque samples were taken at baseline and at 3 months and DNA sequencing was performed for Tanneralla forsythia (T. forsythia), Porphyromonas gingivalis (P. gingivalis), and Treponema denticola (T. denticola).

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy
2. Individuals over 18
3. Periodontitis (4-6 mm pockets) patients with 3 teeth in each half of the jaws except wisdom tooth
4. Non-smoker
5. Not using probiotic tablets/capsules and consuming no more than 3-4 probiotic food.

Exclusion Criteria:

1. Antibiotic use within 6 months.
2. Breastfeeding or pregnancy.
3. Acute oral lesions or necrotizing ulcerative periodontitis
4. Diabetes, rheumatic fever, lung, kidney disease history and drug use that will affect periodontal tissues
5. Patients who smoke or who did not stop until last year
6. Use of probiotics tablets or capsules
7. Probiotic food consumption not more than 3-4 times a week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Periodontal probing depth | Baseline
  the distance from the gingival margin to pocket base.
Periodontal probing depth | 1st month
  the distance from the gingival margin to pocket base.
Periodontal probing depth | 3rd month
  the distance from the gingival margin to pocket base.
Gingival index | Baseline
  It is an index that shows the severity and quantity of gingival inflammation.
Gingival index | 1st month
  It is an index that shows the severity and quantity of gingival inflammation.
Gingival index | 3rd month
  It is an index that shows the severity and quantity of gingival inflammation.
Microbiological sample | Baseline
  Subgingival plaque samples were taken at baseline and at 3 months and DNA sequencing was performed for Tanneralla forsythia, Porphyromonas gingivalis, and Treponema denticola.
Microbiological sample | 1st month
  Subgingival plaque samples were taken at baseline and at 3 months and DNA sequencing was performed for Tanneralla forsythia, Porphyromonas gingivalis, and Treponema denticola.
Microbiological sample | 3rd month
  Subgingival plaque samples were taken at baseline and at 3 months and DNA sequencing was performed for Tanneralla forsythia, Porphyromonas gingivalis, and Treponema denticola.
Plaque index | Baseline
  It is an index that shows the amount of microbial dental plaque on the teeth.
Plaque index | 1st month
  It is an index that shows the amount of microbial dental plaque on the teeth.
Plaque index | 3rd month
  It is an index that shows the amount of microbial dental plaque on the teeth.
Bleeding on probing | Baseline
  Bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus.
Bleeding on probing | 1st month
  Bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus.
Bleeding on probing | 3rd month
  Bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus.

SECONDARY OUTCOMES:
Clinical attachment level | Baseline
  The clinical attachment level is the distance between the enamel-cementum junction and the gingival sulcus.
Clinical attachment level | 1st month
  The clinical attachment level is the distance between the enamel-cementum junction and the gingival sulcus.
Clinical attachment level | 3rd month
  The clinical attachment level is the distance between the enamel-cementum junction and the gingival sulcus.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University Faculty of Dentistry, Ankara
  - Tuğba Şahin, Ankara

IPD SHARING:
Plan to Share IPD: No